CLINICAL TRIAL: NCT04241796
Title: The PATHFINDER Study: Assessment of the Implementation of an Investigational Multi-Cancer Early Detection Test Into Clinical Practice
Brief Title: Assessment of the Implementation of an Investigational Multi-Cancer Early Detection Test Into Clinical Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GRAIL, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GRAIL-007
Record Dates: First submitted 2020-01-02; First posted 2020-01-27 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Elevated Risk and Non-Elevated Risk Groups (Experimental): Two cohorts:
  1. Elevated risk group (approximately 70% of the total enrollment) on the basis of history of smoking, documented genetic cancer predisposition, or personal history of invasive or hematologic malignancy.
  2. Non-elevated risk group (approximately 30% of the total enrollment) with none of the conditions listed in the Elevated Risk Group.
  Interventions: Device: Multi-Cancer Early Detection Test

INTERVENTIONS:
Device: Multi-Cancer Early Detection Test — Blood collection and multi-cancer early detection testing with return of results.

SUMMARY:
PATHFINDER is a prospective, multi-center study in which approximately 6,200 participants will be enrolled. An investigational multi-cancer early detection test, developed by GRAIL, will be ordered by and results returned to a study investigator. In cases with a "signal detected" test result (with a predicted or indeterminate tissue of origin (TOO)), the diagnostic work-up will not be dictated by the protocol, but will instead be coordinated by the ordering and treating medical team at the enrolling sites based on the participant's clinical condition, recommendations by each institution's clinical practices, and in consultation with the study investigator and interdisciplinary care team, as necessary. Additionally, proposed clinical care pathways, developed based on a review of guidelines from the National Comprehensive Cancer Network (NCCN), American College of Radiology (ACR) and other professional organizations, should be referenced by the medical team to determine the diagnostic work-up. The number and types of diagnostic procedures required to achieve diagnostic resolution will be assessed. Performance of multi-cancer early detection test will be evaluated. Additionally, participant-reported outcomes will be collected at several time points to assess participants' perceptions about the multi-cancer early detection test. Participants will be followed for approximately 12 months from the time of enrollment. Cancer status will also be assessed at the 12 month time point.

ELIGIBILITY:
Inclusion Criteria:

Cohort A: Elevated Risk Group (70% of cohort):

* Age: Participant must be 50 years of age or older at the time of signing the Informed Consent Form (ICF).
* Participants must meet at least one of the criteria below:
* History of smoking at least 100 cigarettes in his or her lifetime
* Documented genetic cancer predisposition, hereditary cancer syndrome, or meeting criteria for germline testing based on current NCCN guidelines
* Personal history of invasive or hematologic malignancy, with definitive treatment completed greater than 3 years prior to enrollment. Adjuvant hormone therapy for cancer is permissible (ie may be ongoing within 3 years or at the time of enrollment).

Cohort B: Non-Elevated Risk Group (30% of cohort):

* Age: Participant must be 50 years of age or older, at the time of signing the Informed Consent Form (ICF).
* None of the conditions described in Cohort A, criteria 2a-c
* For all participants, capable of giving signed and legally effective informed consent

Exclusion Criteria:

* Undergoing or referred for diagnostic evaluation due to clinical suspicion for cancer (e.g., referred to a medical or surgical oncologist, or scheduled for biopsy on the basis of a suspicious imaging abnormality).
* Personal history of invasive or hematologic malignancy, diagnosed within the 3 years prior to expected enrollment date, or diagnosed greater than 3 years prior to expected enrollment date and never treated.
* Definitive treatment for invasive or hematologic malignancy within the 3 years prior to expected enrollment date. Adjuvant hormone therapy for cancer is not an exclusion criterion.
* Individuals who will not be able to comply with the protocol procedures.
* Individuals who are not current patients at a participating center.
* Previous or current participation in another GRAIL-sponsored study.
* Previous or current employees or contractors of GRAIL.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6662 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Per participant count of the number and types of diagnostic tests required to achieve diagnostic resolution following a "signal detected" multi-cancer early detection test result. | Until diagnostic resolution or 12 months, whichever occurs first
Per participant time required to achieve diagnostic resolution following a "signal detected" multi-cancer early detection test result. | Until diagnostic resolution or 12 months, whichever occurs first

SECONDARY OUTCOMES:
Positive Predictive Value defined as the proportion of participants with cancer diagnosis out of all participants with "signal detected" multi-cancer early detection test result. | Up to 12 months
Negative Predictive Value defined as the proportion of participants with no cancer diagnosis out of all participants with "signal not detected" results and completed EOS assessment. | Up to 12 months
Specificity defined as the proportion of participants with "signal not detected" results out of all participants with no cancer diagnosis and completed end of study (EOS) assessment. | Up to 12 months
Tissue of origin (TOO) accuracy defined as the proportion of correct TOO predictions in participants with determinate TOO returned by the multi-cancer early detection test and cancer diagnosis. | Up to 12 months
Perceptions of the multi-cancer early detection test result assessed by Adapted Multidimensional Impact of Cancer Risk Assessment (Adapted MICRA). Higher scores represent worse outcomes from 0-95. | Up to 12 months
Changes in health-related quality of life following the multi-cancer early detection test assessed by Short Form Health Survey (SF-12v2). | Up to 12 months
  The SF-12v2 is a measure of health related quality of life. Higher values represent better health e.g. Physical Component Summary (PCS) range from 4.62 to 76.36 and Mental Component Summary (MCS) range from 1.32 to 79.48.
Changes in anxiety following the multi-cancer early detection test result: Patient-reported Outcome Measurement Information System (PROMIS) Anxiety. | Up to 12 months
  Assessed by Patient-reported Outcome Measurement Information System (PROMIS) Anxiety. Range in score from 4 to 20 with higher scores indicate greater severity of anxiety.
Satisfaction with the multi-cancer early detection test: scores | Up to 12 months
  Range in score from 0-100 with higher scores indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Sutter Health, Roseville, California
  - Woodlands Medical Specialists, PA, Pensacola, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - Willamette Valley Cancer Institute, Eugene, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Texas Oncology, PA (West TXO), Amarillo, Texas
  - Intermountain Healthcare Research, St. George, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Northwest Cancer Specialists, P.C. dba Compass Oncology, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nadauld L, McDonnell CH 3rd, Dilaveri CA, Klein EA, Reid R, Marinac CR, Chung KC, Lopatin M, Fung ET, Schrag D, Patrick DL. Psychosocial impact associated with a multicancer early detection test (PATHFINDER): a prospective, multicentre, cohort study. Lancet Oncol. 2025 Feb;26(2):165-174. doi: 10.1016/S1470-2045(24)00645-4. Epub 2025 Jan 13. PMID 39818231
- [Derived] Mahal BA, Margolis M, Hubbell E, Chen C, Venstrom JM, Abran J, Kartlitz JJ, Wyatt AW, Klein EA. A Targeted Methylation-Based Multicancer Early Detection Blood Test Preferentially Detects High-Grade Prostate Cancer While Minimizing Overdiagnosis of Indolent Disease. JCO Precis Oncol. 2024 Aug;8:e2400269. doi: 10.1200/PO.24.00269. PMID 39208374
- [Derived] Schrag D, Beer TM, McDonnell CH 3rd, Nadauld L, Dilaveri CA, Reid R, Marinac CR, Chung KC, Lopatin M, Fung ET, Klein EA. Blood-based tests for multicancer early detection (PATHFINDER): a prospective cohort study. Lancet. 2023 Oct 7;402(10409):1251-1260. doi: 10.1016/S0140-6736(23)01700-2. PMID 37805216